CLINICAL TRIAL: NCT04835831
Title: Interest of APA in Fatty Liver Disease Evaluation of Efficacy and Adherence to an Adapted Physical Activity (APA) Program in Patients With Metabolic Fatty Liver Disease, Open-label, Multicenter, Multicenter Pilot Study
Brief Title: Interest of APA in Fatty Liver Disease Evaluation of Efficacy and Adherence to an Adapted Physical Activity (APA) Program in Patients With Metabolic Fatty Liver Disease
Acronym: STEATO-APA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-AOI-04
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adapted physical activity + Dietetic advice (Experimental)
  Interventions: Other: adapted physical activity + Dietetic advice
- Dietetic advice only (No Intervention)

INTERVENTIONS:
Other: adapted physical activity + Dietetic advice — adapted physical activity during 24 weeks
  Arms: adapted physical activity + Dietetic advice

SUMMARY:
Non-Alcoholic Fatty liver Disease (NAFLD) is a Public Health problem. NAFLD affects nearly 25% of the world's population. NAFLD includes hepatic complications related to insulin resistance and metabolic inflammation. NAFLD is in fact a continuum of liver abnormalities that progresses from pure steatosis, to Non-Alcoholic Steato-Hepatitis-NASH, then to hepatic fibrosis, cirrhosis and even the appearance of primary liver cancer (hepatocellular carcinoma). Although many drugs are being tested for advanced forms of NAFLD, steatohepatitis (NASH) with fibrosis and post-NAFLD cirrhosis, there are currently no drugs with marketing authorization. Excessive and unbalanced dietary intake, excessive physical inactivity and lack of regular physical activity are major contributors to the development of NAFLD. It is therefore logical that the preventive and curative treatment of NAFLD is based on hygienic and dietary measures. Physical exercise alone in patients with NAFLD has been shown to improve liver steatosis even in the absence of weight loss. Proof of concept of the improvement in hepatic steatosis has been shown to be achieved by physical activity, whether or not associated with dietary management. More recently, APA (Adapted Physical Activity) is thus seen as a new modality of care that will become central to the prevention and treatment of NAFLD. The aim of this work is to evaluate the decrease in hepatic steatosis by continuous CAP® and parameters evaluating non-invasive inflammation and hepatic fibrosis in patients with NAFLD subjected to the application of personalized dietary measures without or with the performance of personalized and reproducible physical activity via the prescription of adapted physical activity. The evaluation will be carried out initially, at the end of the operation and 6 months after the end of the operation in order to look for a persistent effect of the modification in lifestyle.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) affects nearly 25% of the world's population and can lead to cirrhosis and hepatocellular carcinoma . Exercise alone in patients with NAFLD has been shown to improve hepatic steatosis. Since 2017, adapted physical activity (APA) has been a medical prescription by the referring physician in France. APA is thus expected to be a new treatment modality that will become central to the prevention and treatment of NAFLD.

The reference examination for the non-invasive quantification of liver steatosis was the Spectro Magnetic Resonance Imaging (MRI) however this technique is expensive and until now reserved for research in highly specialized centers. More recently, the analysis of the MRI signal by a magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) sequence acquired during the performance of a classical MRI scan has been validated as a new, reliable technique that is easier to use routinely than Spectro MRI. However, different technical variants currently not standardized for the quantification of steatosis by PDFF MRI exist. MRI is not widely available and must be performed in a competent and expert center. In contrast, the quantification of steatosis by ultrasound using the classical "Controlled Attenuation Parameter" (CAP®) is available thanks to a FibroScan, which is widely distributed over France. Even if the quantification of steatosis is better by PDFF MRI than by the classical CAP®, the quantification of steatosis by the classical CAP® is well correlated with the hepatic histology.

In addition, several studies have found a decrease in classical CAP® when applying non-drug or drug therapies to lose weight and/or improve insulin resistance in patients with NAFLD. Very recently, Echosens has developed a new technique -the continuous CAP- to improve the reliability of the classical CAP® in the evaluation of steatosis [Audiere et al. ILC 2020]. Continuous CAP® is no longer based on 10 but on 200 measurements of hepatic steatosis. This new measurement technique reduces the variability of the measurement of liver steatosis quantification by 42%.

The aim of this work is to evaluate the decrease in hepatic steatosis by continuous CAP® and parameters evaluating non-invasively inflammation and hepatic fibrosis in patients with NAFLD subjected to the application of personalized dietary measures without or with the performance of personalized and reproducible physical activity via the prescription of an adapted physical activity. The evaluation will be carried out initially, at the end of the APA program and 24 weeks after the end of the APA program in order to look for a persistent effect of the modification in lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Affiliated with social security
* Signature of informed consent
* Diagnosis of NAFLD characterized by the presence of ultrasound steatosis, with a diagnosis made by a physician after a clinical and paraclinical examination as is usually done in routine care and having eliminated another cause of chronic liver disease.
* Effective contraception system for women of childbearing age, a urine pregnancy test will be offered to these women as part of the assessment of the screening visit.

Exclusion Criteria:

* Patient under legal protection
* Refusal to participate in the study
* Alcohol consumption ≥ 30 g/d for men or ≥ 20 g/d for women
* Presence of chronic liver disease from causes other than NAFLDs
* Inability to obtain 10 valid measurements when performing a FibroScan liver elasticity measurement or continuous CAP® steatosis assessment during initial evaluation.
* FibroScan ≥ 20 kPa at initial assessment
* Presence or history of advanced chronic liver disease (cirrhosis) decompensated (Child A6, B or C).
* Known history of a complication related to portal hypertension (including digestive haemorrhage related to portal hypertension, ascites or pleural effusion of cirrhotic cirrhosis, port-pulmonary hypertension).
* Notion of type 2 diabetes unbalanced with an HbA1c ≥ 9%, less than 3 months (measurement of HbA1c is not required before signing the consent form).
* Platelets < 150000/mm3, within the previous 6 months.
* Type 1 diabetes
* Weight loss ≥ 10% of usual body weight, in the 6 months prior to inclusion
* Introduction or dose modification of a GLP1 or orlistat agonist treatment < 1 year
* Practice of regular and/or intense physical activity, weekly (more than 3 hours per week)
* Patients with solid organ or bone marrow transplants
* Patient participating in another study evaluating a therapy to improve non-alcoholic fatty liver disease (NAFLD)
* Contraindication to carrying out APA:

  * Absolute contraindication criteria:

Any unstable pathology affecting a vital organ in particular cardiovascular or pulmonary. Unstable means any situation in which the absence of urgent therapeutic intervention could lead to the death of the patient.

o Contraindication to physical activity Unstable acute coronary syndrome Decompensated heart failure Severe, uncontrolled ventricular rhythm disturbances Presence of an intracardiac thrombus with high embolic risk Presence of a medium to large pericardial effusion Recent history (<6 months) of thrombophlebitis with or without pulmonary embolism Severe and/or symptomatic left ventricular ejection obstruction Any progressive inflammatory and/or infectious disease Severe pulmonary arterial hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Continuous CAP decreased by 10% | evaluated at day 0
  evaluate the decrease in hepatic steatosis by continuous CAP®
Continuous CAP decreased by 10% | evaluated after the 12 weeks
  evaluate the decrease in hepatic steatosis by continuous CAP®

SECONDARY OUTCOMES:
Anthropometric parameters | evaluated at day 0
  assessment of weight
Anthropometric parameters | evaluated after the 12 weeks
  assessment of weight
Muscular performance | evaluated at day 0
  assement with 6-minute walk test
Muscular performance | evaluated after the 12 weeks
  assement with 6-minute walk test
Muscular performance | evaluated after the 24 weeks
  assement with 6-minute walk test
Muscular performance | evaluated after the 48 weeks
  assement with 6-minute walk test
questionnaire: Short Form 36 Health Survey [SF36]. | evaluated at day 0
  assessment between 0 to 100
questionnaire: Short Form 36 Health Survey [SF36]. | evaluated after the 24 weeks
  assessment between 0 to 100
questionnaire: Short Form 36 Health Survey [SF36]. | evaluated after the 48 weeks
  assessment between 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe ANTY, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CHU de Nice, Nice, France
  - Ch de Perpignan, Perpignan, France

IPD SHARING:
Plan to Share IPD: No